CLINICAL TRIAL: NCT04552470
Title: AN 8-WEEK PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF TWICE DAILY PF-06882961 ADMINISTRATION IN JAPANESE ADULTS WITH TYPE 2 DIABETES MELLITUS
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-06882961 in Japanese Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C3421015
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06882961 40 mg (Experimental): Participants will be titrated up to 2 weeks to reach desired dose level
  Interventions: Drug: PF-06882961
- PF-06882961 80 mg (Experimental): Participants will be titrated up to 4 weeks to reach desired dose level
  Interventions: Drug: PF-06882961
- PF-06882961 120 mg (Experimental): Participants will be titrated up to 6 weeks to reach desired dose level
  Interventions: Drug: PF-06882961

INTERVENTIONS:
Drug: Placebo — 3 matching placebo tablets taken twice a day (BID)
  Arms: Placebo
Drug: PF-06882961 — Participants will be randomized to one of 3 active doses (40, 80, or 120 mg), taking 3 tablets twice daily for 8 weeks.
  Arms: PF-06882961 120 mg; PF-06882961 40 mg; PF-06882961 80 mg

SUMMARY:
This is a Phase 1, randomized, double blind (sponsor open), parallel, placebo controlled, twice daily oral dosing study of PF 06882961 in adult Japanese participants with T2DM inadequately controlled on diet and exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who are treated with diet and exercise
* HbA1c greater than or equal to 7% and less than or equal to 10.5%
* Total body weight >50 kg (110 lb) with BMI 22.5 to 45.4 kg/m^2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* Diagnosis of Type 1 diabetes
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, heart failure, or transient ischemic attack within 6 months of screening
* Any malignancy not considered cured
* Personal or family history of MTC or MEN2, or participants with suspected MTC
* Acute pancreatitis or history of chronic pancreatitis
* Symptomatic gallbladder disease
* Known medical history of active proliferative retinopathy and/or macular edema
* Known history of HIV, hepatitis B, hepatitis C or syphilis
* Supine blood pressure greater than or equal to 160 mmHg (systolic) or greater than or equal to 100 mmHg (diastolic)
* Clinically relevant ECG abnormalities
* Positive urine drug test

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one clinic, Keikokai medical corporation, Hachiōji, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 65 participants signed the inform consent form (ICF). 28 participants were screen failures who did not meet criteria and were not enrolled. 37 participants enrolled into the study and assigned to a study treatment.
Groups:
- Placebo: Participants with type 2 diabetes mellitus (T2DM) were randomized to receive placebo matched to PF-06882961 tablet twice daily, for 8 weeks. Post treatment participants were followed approximately for 4 weeks.
- PF-06882961 40 mg: Participants with T2DM were randomized to receive PF-06882961 10 milligram (mg) tablet twice daily on Week 1, 20 mg tablet twice daily on Week 2. After this titration, participants received 40 mg tablet twice daily from Week 3 to 8. Post treatment participants were followed approximately for 4 weeks.
- PF-06882961 80 mg: Participants with T2DM were randomized to receive PF-06882961 10 mg tablet twice daily on Week 1, 20 mg tablet twice daily on Week 2, 40 mg tablet twice daily on Week 3, 60 mg tablet twice daily on Week 4. After this titration, participants received 80 mg tablet twice daily from Week 5 to 8. Post treatment participants were followed approximately for 4 weeks.
- PF-06882961 120 mg: Participants with T2DM were randomized to receive PF-06882961 10 mg tablet twice daily on Week 1, 20 mg tablet twice daily on Week 2, 40 mg tablet twice daily on Week 3, 60 mg tablet twice daily on Week 4, 80 mg tablet twice daily on Week 5, 100 mg tablet twice daily on Week 6. After this titration, participants received 120 mg tablet twice daily from Week 7 to 8. Post treatment participants were followed approximately for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Started | 9 | 10 | 9 | 9
Completed | 9 | 10 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Placebo: Participants with T2DM were randomized to receive placebo matched to PF-06882961 tablet twice daily, for 8 weeks. Post treatment participants were followed approximately for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg | Total
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (8.75) | 55.9 (10.04) | 58.0 (6.69) | 50.7 (7.50) | 55.8 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 5
  Male | 8 | 8 | 8 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 9 | 9 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 10 | 9 | 9 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. Treatment emergent AEs were events between first dose of study drug and approximately 4 weeks after last dose of study drug, that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and all non-serious AEs.
Time Frame: Day 1 of dosing up to approximately 4 weeks after last dose (up to maximum of approximately 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 9 | 10 | 9 | 9
Participants
  Participants with AEs | 3 | 7 | 9 | 9
  Participants with SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Leukocytes (10^9/liter [L]) bilirubin (micromol/L), glucose (millimoles [mmol]/L), triacylglycerol lipase (microkatals [microkat]/L): greater than (>) 1.5*upper limit normal (ULN); activated partial thromboplastin time (s): 1.1*ULN; HDL cholesterol (mmol/L), thyroid stimulating hormone (TSH) (milliunits [mU]/L): less than (<) 0.8*lower limit normal (LLN); LDL cholesterol (mmol/L), urate (mmol/L): >1.2*ULN; triglycerides: >1.3*ULN; aspartate aminotransferase (microkat/L), alanine aminotransferase (microkat/L), gamma glutamyl transferase (microkat/L): >3.0*ULN; cholesterol (mmol/L): >1.3*ULN; urine glucose, ketones urine protein, urine hemoglobin, urobilinogen, nitrite, leukocyte esterase: greater than or equal to (>=) 1; granular casts, hyaline casts: >1.
Time Frame: Day 1 of dosing up to approximately 4 weeks after last dose (up to maximum of approximately 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 9 | 10 | 9 | 9
Participants | 9 | 10 | 8 | 9

3. Primary Outcome: Number of Participants With Absolute Vital Signs (SBP, DBP and Pulse Rate) Values; Increased and Decreased Vital Signs (SBP, DBP) Values From Time-Matched Baseline
Description: Supine systolic blood pressure (SBP) measured in millimeter of mercury (mmHg) had following categories: minimum of absolute SBP <90 mmHg, maximum of SBP >=30 mmHg decrease from baseline and maximum of SBP >=30 mmHg increase from baseline. Supine diastolic blood pressure (DBP) measured in mmHg had following categories: minimum of absolute DBP <50 mmHg, maximum of DBP >20 mmHg decrease from baseline and maximum of DBP >=20 mmHg increase from baseline. Supine pulse rate measured in beats per minute (BPM) had following categories: minimum of absolute supine pulse rate <40 BPM and maximum of absolute supine pulse rate >120 BPM. Baseline was defined as the time-matched value from the average of the triplicate recordings on Day -1.
Time Frame: Baseline (1 Day before dosing) up to last dose (maximum up to Week 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 9 | 10 | 9 | 9
Participants
  Minimum of absolute SBP <90 mmHg | 0 | 0 | 0 | 0
  Maximum of SBP >=30 mmHg decrease | 1 | 0 | 0 | 1
  Maximum of SBP >=30 mmHg increase | 3 | 2 | 3 | 2
  Minimum of absolute DBP <50 mmHg | 0 | 0 | 0 | 0
  Maximum of DBP >=20 mmHg decrease | 0 | 0 | 0 | 0
  Maximum of DBP >=20 mmHg increase | 1 | 2 | 3 | 3
  Minimum of absolute pulse rate <40 BPM | 0 | 0 | 0 | 0
  Maximum of absolute pulse rate >120 BPM | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Absolute Electrocardiogram (ECG) Values and Increased ECG Values From Time-Matched Baseline
Description: PR interval had following categories: maximum absolute PR interval >=300 milliseconds (msec); when baseline PR interval >200 msec and maximum increase from baseline in PR interval >=25 percent; when baseline PR interval less than or equal to (<=) 200 msec and maximum increase from baseline in PR interval >=50 percent. QRS interval had following categories: maximum absolute QRS interval >=140 msec; maximum increase from baseline in QRS interval >=50 percent. QTC interval with Frederica's correction (QTCF) had following categories: absolute QTCF interval >450 msec to <=480 msec; absolute QTCF interval >480 msec to <=500 msec; absolute QTCF interval >500 msec; QTCF interval increase from baseline >=30 msec to <=60 msec; QTCF interval increase from baseline >60 msec.
Time Frame: Baseline (1 Day before dosing) up to last dose (maximum up to Week 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 9 | 10 | 9 | 9
Participants
  Maximum absolute PR >=300 msec | 0 | 0 | 0 | 0
  Baseline PR >200 msec and maximum increase in PR >=25% | 0 | 0 | 0 | 0
  Baseline PR <=200 msec and maximum increase in PR >=50% | 0 | 0 | 0 | 0
  Maximum absolute QRS >=140 msec | 0 | 0 | 0 | 0
  Maximum increase in QRS >=50% | 0 | 0 | 0 | 0
  Absolute QTCF interval >450 msec to <=480 msec | 1 | 0 | 1 | 1
  Absolute QTCF interval >480 msec to <=500 msec | 0 | 0 | 0 | 0
  Absolute QTCF >500 msec | 0 | 0 | 0 | 0
  QTCF increase >=30 msec to <=60 msec | 0 | 0 | 0 | 0
  QTCF increase >60 msec | 0 | 0 | 0 | 0

5. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Zero to Time 24 Hours (AUC24) of PF-06882961
Description: AUC24= Area under the plasma concentration versus time curve from time zero (pre-dose) to time 24 hours (0-24).
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 10, 12, 14 and 24 hours post dose on Day 1 and 56
Population: Pharmacokinetic (PK) parameter analysis set included all participants randomly assigned to study intervention who took at least 1 dose of study intervention and who had at least 1 of the PK parameters of interest calculated. This outcome measure reports AUC24 of PF-06882961, hence there is no data collected and analyzed for reporting arm "Placebo". Here "Number Analyzed" signifies participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 10 | 9 | 9
Nanogram*hour per milliliter
  Day 1 | 414.4 (58) | 500.3 (58) | 484.5 (73)
  Day 56: number analyzed (Participants) | 7 | 6 | 7
  Day 56 | 2424 (45) | 4691 (75) | 6953 (148)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) Observed of PF-06882961
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 10, 12, 14 and 24 hours post dose on Day 1; Pre-dose (0 hour), 1, 2, 4, 6, 8, 10, 12, 14, 24, 36 and 48 hours on Day 56
Population: PK parameter analysis set included all participants randomly assigned to study intervention who took at least 1 dose of study intervention and who had at least 1 of the PK parameters of interest calculated. This outcome measure reports Cmax of PF-06882961, hence there is no data collected and analyzed for reporting arm "Placebo". Here "Number Analyzed" signifies participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 10 | 9 | 9
Nanogram per milliliter
  Day 1 | 32.83 (55) | 45.89 (52) | 39.35 (80)
  Day 56: number analyzed (Participants) | 7 | 6 | 7
  Day 56 | 206.1 (54) | 352.2 (75) | 551.7 (153)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06882961
Time Frame: as for outcome 6
Population: PK parameter analysis set included all participants randomly assigned to study intervention who took at least 1 dose of study intervention and who had at least 1 of the PK parameters of interest calculated. This outcome measure reports Tmax of PF-06882961, hence there is no data collected and analyzed for reporting arm "Placebo". Here "Number Analyzed" signifies participants evaluable at specified time points.
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 10 | 9 | 9
Hours
  Day 1 | 12.0 [2.00 to 23.8] | 12.0 [1.00 to 12.0] | 12.0 [1.00 to 14.0]
  Day 56: number analyzed (Participants) | 7 | 6 | 7
  Day 56 | 12.0 [6.00 to 13.8] | 12.9 [2.00 to 36.0] | 12.0 [0.000 to 13.8]

8. Secondary Outcome: Terminal Phase Half-Life (t1/2) of PF-06882961
Description: t1/2 was calculated as loge (2) per kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 10, 12, 14, 24, 36 and 48 hours on Day 56
Population: PK parameter analysis set included all participants randomly assigned to study intervention who took at least 1 dose of study intervention and who had at least 1 of the PK parameters of interest calculated. This outcome measure reports t1/2 of PF-06882961, hence there is no data collected and analyzed for reporting arm "Placebo".
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
Number analyzed (Participants) | 6 | 3 | 7
Hours | 6.373 (1.7404) | 5.543 (0.30827) | 5.300 (0.80594)

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to approximately 4 weeks after last dose (up to maximum of approximately 12 weeks)
Description: Safety analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Placebo | PF-06882961 40 mg | PF-06882961 80 mg | PF-06882961 120 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 7/10 | 9/9 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | PF-06882961 40 mg (N=10) | PF-06882961 80 mg (N=9) | PF-06882961 120 mg (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4 | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 6 | 8 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5 | 6 | 5
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT04552470/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT04552470/SAP_001.pdf